CLINICAL TRIAL: NCT00136916
Title: Efficacy and Safety of Exubera® (Inhaled Insulin) Compared With Subcutaneous Human Insulin Therapy in Adult Subjects With Type 2 Diabetes Mellitus: A Long-Term, Outpatient, Open-Label, Parallel-Group Comparative Trial
Brief Title: Efficacy and Safety of Inhaled Insulin Compared With Subcutaneous Human Insulin Therapy in Adults With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171029
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exubera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled Insulin (Experimental): Inhalable short-acting insulin
  Interventions: Drug: Inhaled Insulin
- Subcutaneous insulin (Active Comparator)
  Interventions: Drug: Subcutaneous insulin

INTERVENTIONS:
Drug: Inhaled Insulin — Inhaled insulin with dose adjusted according to premeal blood glucose
  Other Names: Exubera
  Arms: Inhaled Insulin
Drug: Subcutaneous insulin — Subcutaneous insulin with dose adjusted according to premeal blood glucose
  Arms: Subcutaneous insulin

SUMMARY:
This study is being done to find out the good and bad effects of inhaled insulin that is used by oral inhalation, to adult males and females with type 2 diabetes mellitus. The other name for this inhaled insulin is Exubera®.

This study included a 2-year comparative treatment period followed by a 6-month follow-up period during which inhaled insulin-treated subjects were switched back to subcutaneous short-acting insulin. After this follow-up period, all eligible subjects entered a comparative extension period that was to last for 5 years. When the comparative portion of the study was terminated, all subjects were requested to return for a final extension follow-up month 3 visit.

DETAILED DESCRIPTION:
Pfizer announced in October 2007 that it would stop marketing Exubera. Nektar, the company from which Pfizer licensed Exubera, announced on April 9, 2008 that it had stopped its search for a new marketing partner. Accordingly, there will be no commercial availability of Exubera. As a result, study A2171029 was terminated on June 9, 2008. Neither safety nor efficacy reasons were the cause of the study termination.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus

Exclusion Criteria:

* COPD
* Asthma
* Smoking Pregnancy

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2002-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (78):
- United States (60):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Luis Obispo, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, Madison, Connecticut
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Chiefland, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Wilmette, Illinois
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Bloomfield Hills, Michigan
  - Pfizer Investigational Site, Plymouth, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Chesterfield, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Mansfield, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (12):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnepeg, Manitoba
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Puerto Rico (4):
  - Pfizer Investigational Site, Aguas Buenas
  - Pfizer Investigational Site, Añasco
  - Pfizer Investigational Site, Cabo Rojo
  - Pfizer Investigational Site, San Juan

REFERENCES:
- [Derived] Rosenstock J, Cefalu WT, Hollander PA, Klioze SS, Reis J, Duggan WT. Safety and efficacy of inhaled human insulin (exubera) during discontinuation and readministration of therapy in adults with type 2 diabetes: a 3-year randomized controlled trial. Diabetes Technol Ther. 2009 Nov;11(11):697-705. doi: 10.1089/dia.2009.0062. PMID 19905885
- [Derived] Rosenstock J, Cefalu WT, Hollander PA, Belanger A, Eliaschewitz FG, Gross JL, Klioze SS, St Aubin LB, Foyt H, Ogawa M, Duggan WT. Two-year pulmonary safety and efficacy of inhaled human insulin (Exubera) in adult patients with type 2 diabetes. Diabetes Care. 2008 Sep;31(9):1723-8. doi: 10.2337/dc08-0159. Epub 2008 Jun 5. PMID 18535196
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171029&StudyName=Efficacy%20and%20Safety%20of%20Inhaled%20Insulin%20Compared%20with%20Subcutaneous%20Human%20Insulin%20Therapy%20in%20Adults%20with%20Type%202%20Diabetes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At screening visit and during the 4-week run-in phase subjects received subcutaneous insulin regime of 2 to 3 daily doses (QD) of regular insulin-/short-acting insulin analog (lispro or aspart) and 1 or 2 doses QD of intermediate or long-acting insulin (neutral protamine hagedorn [NPH] insulin or Ultralente®) or insulin glargine QD at bedtime.
Groups:
- Inhaled Insulin (Exubera®): Pre-prandial inhalable short-acting insulin (INH) regime (packaged as 1 mg and 3 mg inhalation blister packs) plus a single bedtime dose or 2 daily doses of either Ultralene® or NPH insulin, or insulin glargine once daily (QD) at bedtime.
- Subcutaneous Insulin: Subcutaneous (SC) insulin: 2 to 3 daily doses of regular insulin or short-acting insulin analog (lispro or aspart) plus 1 or 2 daily doses of an intermediate to long-acting insulin (NPH insulin or Ultralene®), or insulin glargine QD at bedtime.
Period: Overall Study
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Started | 319 | 316
Received Treatment | 316 | 311
Completed | 194 (At study termination, active subjects completed end-of-study assessment and 3-month follow-up visit) | 212 (At study termination, active subjects completed end-of-study assessment and 3-month follow-up visit)
Not Completed | 125 | 104
Not completed — Never received study treatment | 3 | 5
Not completed — Death | 1 | 3
Not completed — Adverse Event | 27 | 8
Not completed — Laboratory abnormality | 0 | 1
Not completed — Lack of Efficacy | 13 | 3
Not completed — Lost to Follow-up | 12 | 14
Not completed — Withdrawal by Subject | 44 | 46
Not completed — Other | 22 | 24
Not completed — Discontinued in follow up period | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin | Total
Number analyzed (Participants) | 316 | 311 | 627
Age, Customized [Number; unit: participants]
  Between 26 and 35 years | 2 | 7 | 9
  Between 36 and 45 years | 36 | 49 | 85
  Between 46 and 55 years | 100 | 93 | 193
  Between 56 and 65 years | 117 | 101 | 218
  Between 66 and 75 years | 61 | 61 | 122
Age Continuous [Mean (Standard Deviation); unit: years] | 56.7 (9.2) | 55.5 (9.9) | 56.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 118 | 229
  Male | 205 | 193 | 398

OUTCOME MEASURES:

1. Primary Outcome: Change From Month 3 in Forced Expiratory Volume in 1 Second (FEV1)
Description: Change from Month 3: mean of (value of observed FEV1 [forced expiratory volume in the first second of forced exhalation] in liters [L] at treatment observation minus Month 3 value).
Time Frame: Month 3 through extension Month 60
Population: Full analysis set (FAS) FEV1: received at least 1 dose treatment, had baseline and at least 1 post-baseline FEV1. Due to study termination, originally planned inferential analysis for change from Month 3 through extension Month 60 was not done. Cross reference outcome measure: change from baseline in FEV1.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change From Baseline in FEV1
Description: Change from baseline: mean of (value of observed FEV1 [L] at treatment observation minus baseline value).
Time Frame: Baseline through extension follow up Month 3
Population: FAS FEV1; extension Month 36 (M36) Last Observation Carried Forward (LOCF) based on data in the extension phase only; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively. Cross reference outcome measure: change from Month 3 in forced expiratory volume in 1 second.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 311 | 304
L
  Baseline (n=311, 304) | 2.91 (0.68) | 2.93 (0.71)
  Month 3 (M3) (n=290, 291) | -0.06 (0.13) | -0.01 (0.15)
  M6 (n=281, 280) | -0.05 (0.16) | -0.05 (0.17)
  M9 (n=266, 276) | -0.08 (0.17) | -0.07 (0.16)
  M12 (n=259, 263) | -0.09 (0.17) | -0.07 (0.16)
  M15 (n=247, 250) | -0.12 (0.18) | -0.09 (0.17)
  M18 (n=237, 236) | -0.12 (0.18) | -0.10 (0.18)
  M21 (n=232, 233) | -0.13 (0.18) | -0.11 (0.18)
  M24 (n=223, 226) | -0.15 (0.19) | -0.13 (0.18)
  Follow-up (FU) M1 (n=249, 221) | -0.14 (0.18) | -0.14 (0.19)
  FU M3 (n=248, 231) | -0.13 (0.21) | -0.14 (0.20)
  FU M6 (n=242, 220) | -0.12 (0.20) | -0.15 (0.18)
  Extension (Ext) M1 (n=161, 163) | -0.16 (0.20) | -0.16 (0.20)
  Ext M3 (n=157, 158) | -0.19 (0.21) | -0.16 (0.19)
  Ext M6 (n=148, 159) | -0.20 (0.21) | -0.17 (0.20)
  Ext M9 (n=144, 157) | -0.19 (0.21) | -0.16 (0.21)
  Ext M12 (n=144, 157) | -0.20 (0.21) | -0.18 (0.22)
  Ext M15 (n=141, 145) | -0.22 (0.23) | -0.21 (0.20)
  Ext M18 (n=135, 139) | -0.22 (0.23) | -0.21 (0.22)
  Ext M21 (n=132, 143) | -0.23 (0.24) | -0.21 (0.21)
  Ext M24 (n=125, 131) | -0.24 (0.24) | -0.23 (0.22)
  Ext M27 (n=124, 125) | -0.25 (0.23) | -0.24 (0.22)
  Ext M30 (n=125, 126) | -0.24 (0.22) | -0.23 (0.23)
  Ext M33 (n=98, 113) | -0.24 (0.24) | -0.24 (0.22)
  Ext M36 (n=54, 60) | -0.25 (0.18) | -0.28 (0.17)
  Ext M36 [LOCF] (n=171, 169) | -0.24 (0.24) | -0.24 (0.21)
  Ext FU M3 (n=119, 115) | -0.24 (0.21) | -0.25 (0.20)
Statistical Analysis 1: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M3; Test type: Superiority or Other; Mean Difference (Final Values) = -0.045, 90% CI [-0.064 to -0.026], Standard Error of Mean 0.011 — Adjusted Primary Analysis Model includes terms of treatment, baseline pulmonary function tests (PFTs), center, age, sex, and height
Statistical Analysis 2: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M6; Test type: Superiority or Other; Mean Difference (Final Values) = -0.003, 90% CI [-0.025 to 0.020], Standard Error of Mean 0.014 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 3: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M9; Test type: Superiority or Other; Mean Difference (Final Values) = -0.010, 90% CI [-0.033 to 0.013], Standard Error of Mean 0.014 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.020, 90% CI [-0.044 to 0.004], Standard Error of Mean 0.014 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 5: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M15; Test type: Superiority or Other; Mean Difference (Final Values) = -0.023, 90% CI [-0.048 to 0.003], Standard Error of Mean 0.015 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M18; Test type: Superiority or Other; Mean Difference (Final Values) = -0.023, 90% CI [-0.050 to 0.004], Standard Error of Mean 0.016 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M21; Test type: Superiority or Other; Mean Difference (Final Values) = -0.020, 90% CI [-0.047 to 0.007], Standard Error of Mean 0.017 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M24; Test type: Superiority or Other; Mean Difference (Final Values) = -0.026, 90% CI [-0.054 to 0.002], Standard Error of Mean 0.017 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 9: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M1; Test type: Superiority or Other; Mean Difference (Final Values) = 0.007, 90% CI [-0.021 to 0.034], Standard Error of Mean 0.017 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 10: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M3; Test type: Superiority or Other; Mean Difference (Final Values) = 0.014, 90% CI [-0.016 to 0.044], Standard Error of Mean 0.018 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 11: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M6; Test type: Superiority or Other; Mean Difference (Final Values) = 0.027, 90% CI [-0.002 to 0.055], Standard Error of Mean 0.017 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 12: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M1; Test type: Superiority or Other; Mean Difference (Final Values) = -0.004, 90% CI [-0.040 to 0.032], Standard Error of Mean 0.022 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 13: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M3; Test type: Superiority or Other; Mean Difference (Final Values) = -0.033, 90% CI [-0.070 to 0.004], Standard Error of Mean 0.023 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 14: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M6; Test type: Superiority or Other; Mean Difference (Final Values) = -0.039, 90% CI [-0.077 to -0.002], Standard Error of Mean 0.023 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 15: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M9; Test type: Superiority or Other; Mean Difference (Final Values) = -0.036, 90% CI [-0.075 to 0.003], Standard Error of Mean 0.024 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.018, 90% CI [-0.058 to 0.022], Standard Error of Mean 0.024 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 17: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M15; Test type: Superiority or Other; Mean Difference (Final Values) = 0.007, 90% CI [-0.034 to 0.048], Standard Error of Mean 0.025 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M18; Test type: Superiority or Other; Mean Difference (Final Values) = -0.011, 90% CI [-0.055 to 0.033], Standard Error of Mean 0.027 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 19: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M21; Test type: Superiority or Other; Mean Difference (Final Values) = -0.015, 90% CI [-0.058 to 0.029], Standard Error of Mean 0.026 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M24; Test type: Superiority or Other; Mean Difference (Final Values) = -0.015, 90% CI [-0.061 to 0.030], Standard Error of Mean 0.028 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 21: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M27; Test type: Superiority or Other; Mean Difference (Final Values) = -0.000, 90% CI [-0.044 to 0.043], Standard Error of Mean 0.026 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M30; Test type: Superiority or Other; Mean Difference (Final Values) = -0.005, 90% CI [-0.051 to 0.040], Standard Error of Mean 0.027 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 23: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M33; Test type: Superiority or Other; Mean Difference (Final Values) = 0.008, 90% CI [-0.042 to 0.058], Standard Error of Mean 0.030 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M36; Test type: Superiority or Other; Mean Difference (Final Values) = 0.024, 90% CI [-0.030 to 0.077], Standard Error of Mean 0.032 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 25: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M36 LOCF; Test type: Superiority or Other; Mean Difference (Final Values) = -0.003, 90% CI [-0.042 to 0.035], Standard Error of Mean 0.023 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height. Ext M36 (LOCF) based on data in the extension phase only
Statistical Analysis 26: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext FU M3; Test type: Superiority or Other; Mean Difference (Final Values) = 0.019, 90% CI [-0.023 to 0.062], Standard Error of Mean 0.026 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height

3. Primary Outcome: Annual Rate of Change in FEV1
Description: Annual rate of change in FEV1 calculated as slope over time [visit] for forced expiratory volume in 1 second measured as liters per year (L/yr).
Time Frame: Week -2 through extension follow up Month 3 or end of study
Population: FAS FEV1. Due to early termination of study a limited set of analyses were undertaken and results of Annual rate of change in FEV1 were not summarized as planned.
Measure: Mean (Standard Deviation); unit: L/yr
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Summary of ≥ 15 % Decliners in FEV1
Description: Number of subjects with a post-baseline FEV1 decrease of ≥ 15 % [(baseline observed value - visit observed value)/(baseline observed value) * 100]; in the absence of an obvious intercurrrent illness, a repeat FEV1 was performed.
Time Frame: Month 3 through extension follow up Month 3
Population: FAS FEV1; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively.
Measure: Number; unit: participants
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 311 | 304
participants
  M3 (n=290, 291) | 2 | 2
  M6 (n=281, 280) | 3 | 4
  M9 (n=266, 276) | 7 | 5
  M12 (n=259, 263) | 7 | 4
  M15 (n=247, 250) | 13 | 6
  M18 (n=237, 236) | 10 | 8
  M21 (n=232, 233) | 12 | 8
  M24 (n=223, 226) | 14 | 13
  FU M1 (n=249, 221) | 11 | 7
  FU M3 (n=248, 231) | 16 | 15
  FU M6 (n=242, 220) | 13 | 11
  Ext M1 (n=161, 163) | 12 | 6
  Ext M3 (n=157, 158) | 12 | 5
  Ext M6 (n=148, 159) | 14 | 8
  Ext M9 (n=144, 157) | 11 | 10
  Ext M12 (n=144, 157) | 19 | 13
  Ext M15 (n=141, 145) | 15 | 11
  Ext M18 (n=135, 139) | 17 | 18
  Ext M21 (n=132, 143) | 22 | 11
  Ext M24 (n=125, 131) | 22 | 16
  Ext M27 (n=124, 125) | 18 | 14
  Ext M30 (n=125, 126) | 20 | 18
  Ext M33 (n=98, 113) | 10 | 12
  Ext M36 (n=54, 60) | 5 | 6
  Ext FU M3 (n=119, 115) | 14 | 19

5. Primary Outcome: Annual Rate of Change in Carbon Monoxide Diffusion Capacity (DLco)
Description: Annual rate of change in DLco calculated as slope over time (visit) measured as milliliters per minute per millimeters of mercury per year (ml/min/mmHg/yr).
Time Frame: Week -2 through extension follow up Month 3 or end of study
Population: FAS FEV1. Due to early termination of study a limited set of analyses were undertaken and results of Annual rate of change in DLco were not summarized as planned. Cross reference outcome measure: change from baseline in Carbon Monoxide Diffusion Capacity (DLco).
Measure: Mean (Standard Deviation); unit: ml/min/mmHg/yr
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Forced Vital Capacity (FVC) measured in liters (L).
Time Frame: Week -3 through extension follow up Month 3 or end of study
Population: FAS FEV1. Due to early termination of study a limited set of analyses were undertaken and results of FVC were not summarized as planned.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Total Lung Capacity (TLC)
Description: Total Lung Capacity measured in liters (L).
Time Frame: Baseline through extension follow up Month 3
Population: FAS FEV1. Due to early termination of study a limited set of analyses were undertaken and results of TLC were not summarized as planned.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: Change from baseline: mean of (value of observed HbA1c [%] at treatment observation minus baseline value).
Time Frame: Baseline through extension follow up Month 3
Population: FAS HbA1c: received at least 1 dose of study treatment, had baseline HbA1c and at least 1 post-baseline HbA1c; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 315 | 303
percent
  Baseline (n=315, 303) | 7.66 (1.12) | 7.77 (1.12)
  Week 6 (W6) (n=291, 280) | -0.64 (0.67) | -0.60 (0.70)
  M3 (n=296, 291) | -0.80 (0.86) | -0.73 (0.89)
  M6 (n=284, 287) | -0.67 (0.94) | -0.68 (1.00)
  M9 (n=270, 280) | -0.56 (0.98) | -0.61 (0.93)
  M12 (n=261, 263) | -0.45 (0.94) | -0.58 (1.00)
  M15(n=252, 258) | -0.43 (1.00) | -0.51 (1.00)
  M18(n=244, 241) | -0.42 (1.02) | -0.53 (1.06)
  M21 (n=236, 238) | -0.43 (1.04) | -0.52 (1.02)
  M24 (n=226, 234) | -0.35 (1.09) | -0.48 (1.13)
  FU M3 (n=225, 226) | -0.41 (1.04) | -0.44 (1.06)
  FU M6 (n=230, 230) | -0.27 (1.12) | -0.31 (1.06)
  Ext M1 (n=167, 162) | -0.41 (1.16) | -0.40 (1.05)
  Ext M3 (n=164, 162) | -0.33 (1.19) | -0.42 (1.05)
  Ext M6 (n=157, 163) | -0.26 (1.11) | -0.40 (1.10)
  Ext M9 (n=152, 157) | -0.11 (1.15) | -0.26 (1.13)
  Ext M12 (n=150, 157) | -0.08 (1.19) | -0.17 (1.16)
  Ext M15(n=146, 151) | -0.17 (1.30) | -0.25 (1.15)
  Ext M18 (n=145, 145) | -0.20 (1.19) | -0.29 (1.17)
  Ext M21(n=137, 147) | -0.13 (1.16) | -0.20 (1.20)
  Ext M24 (n=131, 137) | -0.18 (1.21) | -0.23 (1.11)
  Ext M27(n=129, 132) | -0.18 (1.13) | -0.28 (1.20)
  Ext M30 (n=129, 129) | -0.20 (1.19) | -0.30 (1.19)
  Ext M33(n=104, 116) | 8.54 (88.44) | -0.18 (1.17)
  Ext M36 (n=55, 64) | -0.20 (1.15) | -0.30 (1.18)
  Ext FU M3 (n=117, 116) | -0.11 (1.40) | -0.17 (1.28)
Statistical Analysis 1: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M3; Test type: Superiority or Other; Mean Difference (Final Values) = -0.119, 90% CI [-0.215 to -0.023], Standard Error of Mean 0.058 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 2: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M6; Test type: Superiority or Other; Mean Difference (Final Values) = -0.023, 90% CI [-0.133 to 0.087], Standard Error of Mean 0.067 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 3: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M9; Test type: Superiority or Other; Mean Difference (Final Values) = 0.010, 90% CI [-0.104 to 0.124], Standard Error of Mean 0.069 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 4: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M12; Test type: Superiority or Other; Mean Difference (Final Values) = 0.091, 90% CI [-0.033 to 0.214], Standard Error of Mean 0.075 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 5: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M15; Test type: Superiority or Other; Mean Difference (Final Values) = 0.052, 90% CI [-0.081 to 0.185], Standard Error of Mean 0.081 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 6: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M18; Test type: Superiority or Other; Mean Difference (Final Values) = 0.090, 90% CI [-0.054 to 0.234], Standard Error of Mean 0.087 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 7: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M21; Test type: Superiority or Other; Mean Difference (Final Values) = 0.068, 90% CI [-0.073 to 0.208], Standard Error of Mean 0.085 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 8: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M24; Test type: Superiority or Other; Mean Difference (Final Values) = 0.100, 90% CI [-0.058 to 0.257], Standard Error of Mean 0.096 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 9: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M3; Test type: Superiority or Other; Mean Difference (Final Values) = 0.006, 90% CI [-0.143 to 0.154], Standard Error of Mean 0.090 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 10: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M6; Test type: Superiority or Other; Mean Difference (Final Values) = 0.036, 90% CI [-0.119 to 0.190], Standard Error of Mean 0.094 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 11: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M1; Test type: Superiority or Other; Mean Difference (Final Values) = -0.019, 90% CI [-0.200 to 0.161], Standard Error of Mean 0.110 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 12: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M3; Test type: Superiority or Other; Mean Difference (Final Values) = 0.081, 90% CI [-0.101 to 0.263], Standard Error of Mean 0.110 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 13: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M6; Test type: Superiority or Other; Mean Difference (Final Values) = 0.141, 90% CI [-0.038 to 0.320], Standard Error of Mean 0.108 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 14: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M9; Test type: Superiority or Other; Mean Difference (Final Values) = 0.150, 90% CI [-0.041 to 0.342], Standard Error of Mean 0.116 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 15: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M12; Test type: Superiority or Other; Mean Difference (Final Values) = 0.104, 90% CI [-0.090 to 0.298], Standard Error of Mean 0.118 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 16: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M15; Test type: Superiority or Other; Mean Difference (Final Values) = 0.074, 90% CI [-0.132 to 0.279], Standard Error of Mean 0.125 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 17: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M18; Test type: Superiority or Other; Mean Difference (Final Values) = 0.087, 90% CI [-0.111 to 0.284], Standard Error of Mean 0.120 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 18: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M21; Test type: Superiority or Other; Mean Difference (Final Values) = 0.064, 90% CI [-0.141 to 0.270], Standard Error of Mean 0.124 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 19: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M24; Test type: Superiority or Other; Mean Difference (Final Values) = 0.047, 90% CI [-0.156 to 0.249], Standard Error of Mean 0.123 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 20: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M27; Test type: Superiority or Other; Mean Difference (Final Values) = 0.067, 90% CI [-0.138 to 0.272], Standard Error of Mean 0.124 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 21: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M30; Test type: Superiority or Other; Mean Difference (Final Values) = 0.046, 90% CI [-0.171 to 0.264], Standard Error of Mean 0.132 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 22: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M33; Test type: Superiority or Other; Mean Difference (Final Values) = 9.824, 90% CI [-3.920 to 23.569], Standard Error of Mean 8.319 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 23: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M36; Test type: Superiority or Other; Mean Difference (Final Values) = 0.011, 90% CI [-0.316 to 0.337], Standard Error of Mean 0.197 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center
Statistical Analysis 24: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext FU M3; Test type: Superiority or Other; Mean Difference (Final Values) = 0.024, 90% CI [-0.245 to 0.292], Standard Error of Mean 0.163 — Adjusted Primary Analysis Model includes terms of treatment, baseline HbA1c, and center

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline: mean of (value of observed FPG [milligrams per deciliter (mg/dL)] at treatment observation minus baseline value).
Time Frame: Baseline through extension follow up Month 3
Population: FAS HbA1c; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 315 | 303
mg/dL
  Baseline (n=315, 303) | 158.13 (42.71) | 154.53 (41.51)
  W6 (n=282, 276) | -23.36 (51.69) | -12.55 (50.46)
  M3 (n=294, 290) | -26.38 (52.72) | -12.77 (54.93)
  M6 (n=281, 285) | -25.21 (53.48) | -9.05 (68.42)
  M9 (n=267, 279) | -26.68 (54.95) | -10.41 (56.42)
  M12 (n=260, 263) | -20.55 (59.68) | -7.60 (60.03)
  M15(n=253, 255) | -21.37 (54.53) | -8.82 (55.57)
  M18(n=242, 238) | -24.52 (54.50) | -7.69 (58.47)
  M21(n=232, 237) | -25.95 (53.06) | -13.14 (54.66)
  M24 (n=226, 232) | -24.02 (54.45) | -8.91 (65.24)
  FU M3 (n=5, 4) | -22.60 (44.65) | -4.08 (32.08)
  FU M6 (n=161, 156) | -2.85 (66.18) | -1.56 (71.72)
  Ext M1 (n=165, 162) | -17.91 (60.96) | -7.34 (60.98)
  Ext M3 (n=162, 159) | -18.16 (66.59) | -9.29 (62.50)
  Ext M6 (n=152, 161) | -15.65 (67.18) | -4.34 (61.96)
  Ext M9 (n=149, 155) | -13.99 (61.68) | -6.06 (60.86)
  Ext M12 (n=148, 155) | -12.53 (72.25) | -4.98 (62.92)
  Ext M15(n=143, 143) | -6.88 (68.85) | -4.23 (65.21)
  Ext M18 (n=136, 138) | -17.23 (65.97) | -10.32 (63.11)
  Ext M21(n=132, 144) | -12.86 (63.98) | -6.53 (64.09)
  Ext M24 (n=129, 136) | -14.45 (61.65) | -3.47 (68.57)
  Ext M27 (n=128, 129) | -21.68 (58.35) | -3.76 (63.31)
  Ext M30 (n=127, 130) | -11.80 (62.82) | -6.40 (61.47)
  Ext M33(n=103, 115) | -16.26 (63.44) | -7.35 (66.21)
  Ext M36 (n=55, 64) | -28.61 (65.99) | -13.35 (53.97)
  Ext FU M3 (n=115, 118) | -2.87 (81.19) | 1.88 (64.94)
Statistical Analysis 1: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M3; Test type: Superiority or Other; Mean Difference (Final Values) = -12.39, 90% CI [-19.07 to -5.710], Standard Error of Mean 4.054 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 2: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M6; Test type: Superiority or Other; Mean Difference (Final Values) = -14.21, 90% CI [-22.11 to -6.312], Standard Error of Mean 4.795 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 3: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M12; Test type: Superiority or Other; Mean Difference (Final Values) = -10.96, 90% CI [-19.07 to -2.852], Standard Error of Mean 4.920 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 4: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M24; Test type: Superiority or Other; Mean Difference (Final Values) = -12.56, 90% CI [-20.89 to -4.232], Standard Error of Mean 5.052 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 5: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M3; Test type: Superiority or Other; Mean Difference (Final Values) = -16.83, 90% CI [-80.69 to 47.019], Standard Error of Mean 21.867 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 6: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M6; Test type: Superiority or Other; Mean Difference (Final Values) = 2.578, 90% CI [-9.257 to 14.412], Standard Error of Mean 7.173 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 7: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M1; Test type: Superiority or Other; Mean Difference (Final Values) = -9.460, 90% CI [-19.37 to 0.450], Standard Error of Mean 6.007 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 8: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M3; Test type: Superiority or Other; Mean Difference (Final Values) = -9.481, 90% CI [-20.11 to 1.153], Standard Error of Mean 6.446 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 9: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M6; Test type: Superiority or Other; Mean Difference (Final Values) = -10.76, 90% CI [-21.95 to 0.438], Standard Error of Mean 6.785 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 10: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M9; Test type: Superiority or Other; Mean Difference (Final Values) = -6.827, 90% CI [-16.98 to 3.328], Standard Error of Mean 6.154 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 11: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M12; Test type: Superiority or Other; Mean Difference (Final Values) = -7.287, 90% CI [-19.15 to 4.579], Standard Error of Mean 7.192 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 12: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M15; Test type: Superiority or Other; Mean Difference (Final Values) = -1.848, 90% CI [-13.76 to 10.066], Standard Error of Mean 7.219 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 13: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M18; Test type: Superiority or Other; Mean Difference (Final Values) = -9.022, 90% CI [-20.83 to 2.790], Standard Error of Mean 7.156 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 14: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M21; Test type: Superiority or Other; Mean Difference (Final Values) = -7.078, 90% CI [-18.99 to 4.834], Standard Error of Mean 7.217 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 15: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M24; Test type: Superiority or Other; Mean Difference (Final Values) = -12.53, 90% CI [-24.63 to -0.429], Standard Error of Mean 7.329 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 16: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M27; Test type: Superiority or Other; Mean Difference (Final Values) = -19.07, 90% CI [-30.45 to -7.685], Standard Error of Mean 6.895 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 17: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M30; Test type: Superiority or Other; Mean Difference (Final Values) = -3.220, 90% CI [-15.15 to 8.705], Standard Error of Mean 7.223 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 18: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M33; Test type: Superiority or Other; Mean Difference (Final Values) = -8.490, 90% CI [-21.09 to 4.107], Standard Error of Mean 7.625 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 19: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M36; Test type: Superiority or Other; Mean Difference (Final Values) = -21.88, 90% CI [-36.66 to -7.105], Standard Error of Mean 8.906 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center
Statistical Analysis 20: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext FU M3; Test type: Superiority or Other; Mean Difference (Final Values) = -4.673, 90% CI [-19.16 to 9.812], Standard Error of Mean 8.770 — Adjusted Primary Analysis Model includes terms of treatment, baseline fasting plasma glucose, and center

10. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline: mean of (value of observed body weight [kilograms (kg)] at treatment observation minus baseline value).
Time Frame: Baseline through extension follow up Month 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 314 | 302
kg
  Baseline (n=314, 302) | 87.18 (14.75) | 88.31 (15.50)
  W4 (n=280, 270) | 0.63 (2.11) | 0.83 (1.86)
  W8 (n=289, 281) | 1.07 (2.41) | 1.00 (2.31)
  M3 (n=288, 290) | 1.08 (2.75) | 1.13 (2.55)
  W18(n=280, 285) | 1.33 (3.13) | 1.76 (3.03)
  M6 (n=276, 277) | 1.15 (3.59) | 1.89 (3.53)
  M9 (n=269, 274) | 1.50 (3.95) | 2.15 (3.90)
  M12 (n=259, 264) | 1.75 (4.29) | 2.37 (4.34)
  M15(n=247, 249) | 1.88 (4.33) | 2.62 (4.49)
  M18(n=237, 235) | 1.79 (4.53) | 2.93 (4.85)
  M21(n=232, 232) | 1.99 (4.56) | 3.04 (5.04)
  M24 (n=223, 226) | 2.04 (4.86) | 3.36 (5.16)
  FU M3 (n=249, 231) | 2.32 (5.25) | 3.63 (5.34)
  FU M6 (n=243, 218) | 2.38 (5.34) | 4.09 (7.70)
  Ext M1 (n=161, 162) | 2.87 (5.48) | 3.75 (5.58)
  Ext M3 (n=157, 157) | 2.83 (4.78) | 4.14 (5.69)
  Ext M6 (n=148, 159) | 3.15 (5.70) | 4.01 (6.07)
  Ext M9 (n=144, 156) | 2.95 (5.95) | 3.89 (5.87)
  Ext M12 (n=144, 156) | 2.96 (6.00) | 4.19 (6.12)
  Ext M15 (n=142, 145) | 3.12 (5.91) | 4.54 (6.26)
  Ext M18 (n=135, 139) | 3.33 (9.20) | 4.46 (6.12)
  Ext M21(n=132, 143) | 2.79 (6.90) | 5.01 (8.37)
  Ext M24 (n=126, 131) | 2.94 (6.98) | 4.57 (6.37)
  Ext M27(n=125, 125) | 2.99 (6.94) | 5.58 (9.62)
  Ext M30 (n=125, 126) | 3.39 (6.43) | 4.78 (6.96)
  Ext M33(n=99, 113) | 2.77 (6.33) | 5.22 (7.21)
  Ext M36 (n=54, 60) | 2.48 (6.61) | 5.28 (7.09)
  Ext FU M3 (n=119, 115) | 2.74 (6.90) | 4.44 (6.87)
Statistical Analysis 1: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M3; Test type: Superiority or Other; Mean Difference (Final Values) = -0.059, 90% CI [-0.416 to 0.299], Standard Error of Mean 0.217 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 2: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M6; Test type: Superiority or Other; Mean Difference (Final Values) = -0.735, 90% CI [-1.224 to -0.246], Standard Error of Mean 0.297 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 3: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.642, 90% CI [-1.251 to -0.032], Standard Error of Mean 0.370 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 4: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M24; Test type: Superiority or Other; Mean Difference (Final Values) = -1.355, 90% CI [-2.120 to -0.589], Standard Error of Mean 0.464 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 5: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M3; Test type: Superiority or Other; Mean Difference (Final Values) = -1.303, 90% CI [-2.086 to -0.520], Standard Error of Mean 0.475 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 6: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M6; Test type: Superiority or Other; Mean Difference (Final Values) = -1.557, 90% CI [-2.539 to -0.575], Standard Error of Mean 0.596 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 7: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M1; Test type: Superiority or Other; Mean Difference (Final Values) = -0.904, 90% CI [-1.898 to 0.090], Standard Error of Mean 0.603 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 8: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M3; Test type: Superiority or Other; Mean Difference (Final Values) = -1.280, 90% CI [-2.225 to -0.334], Standard Error of Mean 0.573 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 9: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M6; Test type: Superiority or Other; Mean Difference (Final Values) = -0.834, 90% CI [-1.909 to 0.241], Standard Error of Mean 0.652 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 10: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M9; Test type: Superiority or Other; Mean Difference (Final Values) = -1.001, 90% CI [-2.080 to 0.078], Standard Error of Mean 0.654 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 11: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M12; Test type: Superiority or Other; Mean Difference (Final Values) = -1.316, 90% CI [-2.431 to -0.200], Standard Error of Mean 0.676 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 12: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M15; Test type: Superiority or Other; Mean Difference (Final Values) = -1.512, 90% CI [-2.661 to -0.363], Standard Error of Mean 0.696 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 13: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M18; Test type: Superiority or Other; Mean Difference (Final Values) = -1.313, 90% CI [-2.824 to 0.198], Standard Error of Mean 0.916 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 14: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M21; Test type: Superiority or Other; Mean Difference (Final Values) = -2.399, 90% CI [-3.891 to -0.907], Standard Error of Mean 0.904 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 15: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M24; Test type: Superiority or Other; Mean Difference (Final Values) = -1.566, 90% CI [-2.867 to -0.265], Standard Error of Mean 0.788 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 16: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M27; Test type: Superiority or Other; Mean Difference (Final Values) = -2.720, 90% CI [-4.439 to -1.001], Standard Error of Mean 1.041 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 17: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M30; Test type: Superiority or Other; Mean Difference (Final Values) = -1.401, 90% CI [-2.755 to -0.047], Standard Error of Mean 0.820 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 18: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M33; Test type: Superiority or Other; Mean Difference (Final Values) = -2.281, 90% CI [-3.781 to -0.782], Standard Error of Mean 0.908 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 19: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M36; Test type: Superiority or Other; Mean Difference (Final Values) = -2.766, 90% CI [-4.932 to -0.599], Standard Error of Mean 1.305 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center
Statistical Analysis 20: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext FU M3; Test type: Superiority or Other; Mean Difference (Final Values) = -1.637, 90% CI [-3.120 to -0.153], Standard Error of Mean 0.898 — Adjusted Primary Analysis Model includes terms of treatment, baseline weight, and center

11. Secondary Outcome: Total Daily Long-acting Insulin Dose (Unadjusted for Body Weight)
Description: Total daily long-acting insulin dose unadjusted for body weight. Long-acting (units) insulin for inhaled insulin and subcutaneous treatment groups included NPH insulin, Ultralente®, and insulin glargine.
Time Frame: Month 3 through extension Month 36
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 315 | 303
units
  M3 (n=301, 298) | 44.10 (25.60) | 47.98 (25.06)
  M6 (n=289, 291) | 44.03 (26.27) | 47.31 (25.47)
  M9 (n=275, 284) | 43.64 (26.17) | 48.11 (26.02)
  M12 (n=266, 270) | 44.62 (27.43) | 48.01 (26.02)
  M15 (n=258, 260) | 45.02 (27.76) | 48.37 (26.48)
  M18 (n=243, 242) | 46.07 (27.77) | 48.93 (27.60)
  M21 (n=240, 240) | 46.67 (29.06) | 49.84 (28.73)
  M24 (n=229, 237) | 46.62 (28.55) | 50.34 (29.31)
  Ext M1 (n=167, 164) | 45.29 (28.00) | 51.29 (28.45)
  Ext M3 (n=165, 162) | 45.76 (28.61) | 51.62 (28.71)
  Ext M6 (n=159, 164) | 45.89 (28.61) | 52.18 (28.85)
  Ext M9 (n=156, 158) | 46.51 (29.34) | 52.32 (28.89)
  Ext M12 (n=151, 158) | 46.52 (29.84) | 51.72 (29.06)
  Ext M15 (n=148, 149) | 46.39 (30.12) | 52.92 (29.83)
  Ext M18 (n=145, 145) | 46.31 (31.17) | 52.37 (29.78)
  Ext M21 (n=137, 148) | 46.49 (31.17) | 52.68 (29.40)
  Ext M24 (n=131, 137) | 47.21 (32.42) | 52.18 (30.33)
  Ext M27 (n=132, 133) | 48.13 (32.76) | 52.42 (29.87)
  Ext M30 (n=131, 130) | 48.13 (33.41) | 53.22 (29.85)
  Ext M33 (n=104, 116) | 48.38 (32.47) | 51.93 (30.65)
  Ext M36 (n=56, 65) | 46.42 (31.91) | 53.47 (28.96)

12. Secondary Outcome: Total Daily Long-acting Insulin (Adjusted for Body Weight)
Description: Total daily dose of long-acting insulin adjusted for body weight (units per kilogram [kg]). Long-acting (units) insulin for inhaled insulin and subcutaneous treatment groups included NPH insulin, Ultralente®, and insulin glargine.
Time Frame: Month 3 through extension Month 36
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 315 | 303
units/kg
  M3 (n=301, 298) | 0.51 (0.29) | 0.54 (0.27)
  M6 (n=289, 291) | 0.50 (0.29) | 0.54 (0.28)
  M9 (n=275, 284) | 0.50 (0.29) | 0.55 (0.29)
  M12 (n=266, 270) | 0.51 (0.30) | 0.55 (0.29)
  M15 (n=258, 260) | 0.52 (0.31) | 0.56 (0.30)
  M18 (n=243, 242) | 0.53 (0.31) | 0.57 (0.31)
  M21 (n=240, 240) | 0.53 (0.32) | 0.57 (0.32)
  M24 (n=229, 237) | 0.54 (0.32) | 0.58 (0.32)
  Ext M1 (n=167, 164) | 0.53 (0.33) | 0.59 (0.31)
  Ext M3 (n=165, 162) | 0.53 (0.34) | 0.59 (0.31)
  Ext M6 (n=159, 164) | 0.54 (0.34) | 0.60 (0.31)
  Ext M9 (n=156, 158) | 0.54 (0.35) | 0.60 (0.31)
  Ext M12 (n=151, 158) | 0.54 (0.36) | 0.60 (0.32)
  Ext M15 (n=148, 149) | 0.54 (0.36) | 0.61 (0.32)
  Ext M18 (n=145, 145) | 0.54 (0.37) | 0.61 (0.32)
  Ext M21 (n=137, 148) | 0.54 (0.37) | 0.61 (0.32)
  Ext M24 (n=131, 137) | 0.55 (0.39) | 0.61 (0.34)
  Ext M27 (n=132, 133) | 0.56 (0.39) | 0.61 (0.33)
  Ext M30 (n=131, 130) | 0.56 (0.41) | 0.62 (0.33)
  Ext M33 (n=104, 116) | 0.56 (0.37) | 0.61 (0.34)
  Ext M36 (n=56, 65) | 0.53 (0.37) | 0.61 (0.31)

13. Secondary Outcome: Total Daily Short-acting Insulin Dose (Unadjusted for Body Weight)
Description: Total daily dose of short-acting insulin unadjusted for body weight. Short-acting insulin (milligrams [mg]) for the inhaled insulin treatment group was inhaled insulin; short-acting insulin (units) for the subcutaneous insulin treatment group included insulin lispro, insulin aspart, and regular insulin.
Time Frame: Month 3 through extension Month 36
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg, units
Groups:
- Inhaled Insulin (Exubera®) (mg): Pre-prandial inhalable short-acting insulin (INH) regime (packaged as 1 mg and 3 mg inhalation blister packs) plus a single bedtime dose or 2 daily doses of either Ultralene® or NPH insulin, or insulin glargine once daily (QD) at bedtime.
- Subcutaneous Insulin (Units): Subcutaneous (SC) insulin: 2 to 3 daily doses of regular insulin or short-acting insulin analog (lispro or aspart) plus 1 or 2 daily doses of an intermediate to long-acting insulin (NPH insulin or Ultralene®), or insulin glargine QD at bedtime.
Arm/Group | Inhaled Insulin (Exubera®) (mg) | Subcutaneous Insulin (Units)
Number analyzed (Participants) | 315 | 303
mg, units
  M3 (n=302, 299) | 12.66 (6.80) | 31.15 (18.75)
  M6 (n=290, 292) | 13.18 (6.90) | 31.73 (19.08)
  M9 (n=275, 285) | 13.57 (7.57) | 31.58 (18.89)
  M12 (n=266, 270) | 14.40 (7.90) | 31.94 (19.29)
  M15 (n=258, 261) | 14.70 (8.06) | 31.88 (19.37)
  M18 (n=245, 242) | 14.91 (8.41) | 32.79 (20.70)
  M21 (n=240, 242) | 15.09 (8.55) | 33.18 (20.92)
  M24 (n=229, 238) | 15.43 (8.65) | 34.04 (21.84)
  Ext M1 (n=167, 164) | 13.89 (8.47) | 34.52 (24.52)
  Ext M3 (n=165, 163) | 14.62 (9.18) | 35.29 (23.19)
  Ext M6 (n=159, 165) | 14.62 (9.16) | 35.43 (24.80)
  Ext M9 (n=156, 161) | 14.82 (9.10) | 35.68 (24.72)
  Ext M12 (n=151, 160) | 15.42 (9.81) | 36.56 (26.34)
  Ext M15 (n=148, 151) | 15.48 (9.90) | 36.27 (25.51)
  Ext M18 (n=145, 146) | 15.57 (9.93) | 37.37 (26.29)
  Ext M21 (n=138, 149) | 15.94 (10.41) | 36.80 (27.09)
  Ext M24 (n=131, 138) | 15.46 (9.70) | 38.51 (29.06)
  Ext M27 (n=132, 134) | 16.25 (10.30) | 38.54 (28.13)
  Ext M30 (n=131, 131) | 16.56 (10.63) | 39.01 (28.66)
  Ext M33 (n=105, 117) | 16.51 (10.43) | 40.33 (30.81)
  Ext M36 (n=56, 66) | 17.25 (11.30) | 42.34 (28.72)

14. Secondary Outcome: Total Daily Short-acting Insulin Dose (Adjusted for Body Weight)
Description: Total daily dose of short-acting insulin adjusted for body weight. Short-acting insulin (mg) for the inhaled insulin treatment group was inhaled insulin (mg divided by kg); short-acting insulin (units) for the subcutaneous insulin treatment group included insulin lispro, insulin aspart, and regular insulin (units divided by kg).
Time Frame: Month 3 through extension Month 36
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/kg, units/kg
Arm/Group | Inhaled Insulin (Exubera®) (mg) | Subcutaneous Insulin (Units)
Number analyzed (Participants) | 315 | 303
mg/kg, units/kg
  M3 (n=302, 299) | 0.15 (0.07) | 0.36 (0.22)
  M6 (n=290, 292) | 0.15 (0.08) | 0.36 (0.22)
  M9 (n=275, 285) | 0.16 (0.08) | 0.36 (0.22)
  M12 (n=266, 270) | 0.17 (0.09) | 0.37 (0.23)
  M15 (n=258, 261) | 0.17 (0.09) | 0.37 (0.24)
  M18 (n=245, 242) | 0.17 (0.09) | 0.38 (0.25)
  M21 (n=240, 242) | 0.17 (0.09) | 0.39 (0.26)
  M24 (n=229, 238) | 0.18 (0.10) | 0.40 (0.27)
  Ext M1 (n=167, 164) | 0.16 (0.09) | 0.40 (0.30)
  Ext M3 (n=165, 163) | 0.17 (0.10) | 0.41 (0.26)
  Ext M6 (n=159, 165) | 0.17 (0.10) | 0.41 (0.30)
  Ext M9 (n=156, 161) | 0.17 (0.10) | 0.42 (0.30)
  Ext M12 (n=151, 160) | 0.18 (0.11) | 0.43 (0.32)
  Ext M15 (n=148, 151) | 0.18 (0.11) | 0.42 (0.31)
  Ext M18 (n=145, 146) | 0.18 (0.11) | 0.44 (0.32)
  Ext M21 (n=138, 149) | 0.18 (0.11) | 0.43 (0.33)
  Ext M24 (n=131, 138) | 0.18 (0.10) | 0.45 (0.35)
  Ext M27 (n=132, 134) | 0.19 (0.11) | 0.45 (0.34)
  Ext M30 (n=131, 131) | 0.19 (0.12) | 0.46 (0.34)
  Ext M33 (n=105, 117) | 0.19 (0.11) | 0.47 (0.36)
  Ext M36 (n=56, 66) | 0.19 (0.12) | 0.48 (0.31)

15. Secondary Outcome: Lipid Panel: Total Cholesterol, High Density Lipoprotein, Low Density Lipoprotein, and Triglycerides
Description: Lipid values for total cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL), and triglycerides measured as milligrams per deciliter (mg/dL).
Time Frame: Week -4 through Month 24
Population: FAS: received at least 1 dose of study treatment. Due to early termination of study a limited set of analyses were undertaken and results of Lipids were not summarized as planned.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Change From Baseline in Carbon Monoxide Diffusion Capacity (DLco)
Description: Change from baseline: mean of (value of observed DLco [milliliters per minute per millimeters of mercury (ml/min/mmHg)] at treatment observation minus baseline value).
Time Frame: Baseline through extension follow up Month 3
Population: FAS FEV1; extension M36 LOCF based on data in the extension phase only; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively. Cross reference outcome measure Annual rate of change in Carbon Monoxide Diffusion Capacity (DLco).
Measure: Mean (Standard Deviation); unit: ml/min/mmHg
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 308 | 303
ml/min/mmHg
  Baseline (n=308, 303) | 24.13 (5.54) | 23.97 (5.72)
  M3 (n=289, 290) | -0.57 (1.60) | -0.32 (1.62)
  M6 (n=278, 280) | -0.56 (1.62) | -0.44 (1.73)
  M9 (n=266, 272) | -0.67 (1.78) | -0.72 (1.77)
  M12 (n=258, 263) | -0.72 (1.86) | -0.41 (1.87)
  M15 (n=246, 248) | -0.81 (1.83) | -0.56 (1.96)
  M18 (n=237, 232) | -0.86 (1.95) | -0.65 (1.92)
  M21 (n=231, 231) | -0.89 (1.98) | -0.67 (1.92)
  M24 (n=221, 223) | -0.74 (2.10) | -0.81 (2.06)
  FU M1 (n=247, 220) | -0.46 (2.05) | -1.02 (2.01)
  FU M3 (n=247, 231) | -0.58 (2.07) | -0.90 (2.15)
  FU M6 (n=241, 219) | -0.64 (2.15) | -0.95 (2.11)
  Ext M1 (n=159, 161) | -1.01 (2.08) | -1.09 (2.15)
  Ext M3 (n=157, 157) | -1.07 (2.10) | -1.16 (2.45)
  Ext M6 (n=148, 157) | -1.48 (1.87) | -1.26 (2.38)
  Ext M9 (n=143, 155) | -1.15 (2.31) | -1.36 (2.54)
  Ext M12 (n=141, 155) | -1.49 (2.22) | -1.59 (2.38)
  Ext M15 (n=141, 142) | -1.49 (2.25) | -1.46 (2.41)
  Ext M18 (n=132, 138) | -1.54 (2.25) | -1.63 (2.21)
  Ext M21 (n=129, 142) | -1.33 (2.45) | -1.64 (2.45)
  Ext M24 (n=124, 130) | -1.39 (2.27) | -1.46 (2.43)
  Ext M27 (n=123, 124) | -1.35 (2.48) | -1.44 (2.41)
  Ext M30 (n=124, 125) | -1.75 (2.13) | -1.62 (2.55)
  Ext M33 (n=98, 113) | -1.47 (2.05) | -1.61 (2.25)
  Ext M36 (n=52, 60) | -1.22 (2.16) | -1.87 (2.23)
  Ext M36 [LOCF] (n=171, 169) | -1.39 (2.31) | -1.77 (2.46)
  Ext FU M3 (n=118, 114) | -1.12 (2.15) | -1.69 (2.56)
Statistical Analysis 1: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M3; Test type: Superiority or Other; Mean Difference (Final Values) = -0.251, 90% CI [-0.466 to -0.037], Standard Error of Mean 0.130 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 2: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M6; Test type: Superiority or Other; Mean Difference (Final Values) = -0.095, 90% CI [-0.323 to 0.134], Standard Error of Mean 0.139 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 3: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M9; Test type: Superiority or Other; Mean Difference (Final Values) = 0.084, 90% CI [-0.158 to 0.325], Standard Error of Mean 0.146 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 4: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.266, 90% CI [-0.524 to -0.009], Standard Error of Mean 0.156 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 5: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M15; Test type: Superiority or Other; Mean Difference (Final Values) = -0.181, 90% CI [-0.453 to 0.091], Standard Error of Mean 0.165 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 6: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M18; Test type: Superiority or Other; Mean Difference (Final Values) = -0.141, 90% CI [-0.427 to 0.145], Standard Error of Mean 0.173 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 7: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M21; Test type: Superiority or Other; Mean Difference (Final Values) = -0.155, 90% CI [-0.445 to 0.134], Standard Error of Mean 0.176 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 8: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; M24; Test type: Superiority or Other; Mean Difference (Final Values) = 0.119, 90% CI [-0.193 to 0.431], Standard Error of Mean 0.189 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 9: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M1; Test type: Superiority or Other; Mean Difference (Final Values) = 0.617, 90% CI [0.322 to 0.911], Standard Error of Mean 0.179 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 10: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M3; Test type: Superiority or Other; Mean Difference (Final Values) = 0.354, 90% CI [0.051 to 0.657], Standard Error of Mean 0.184 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 11: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; FU M6; Test type: Superiority or Other; Mean Difference (Final Values) = 0.318, 90% CI [0.011 to 0.626], Standard Error of Mean 0.186 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 12: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M1; Test type: Superiority or Other; Mean Difference (Final Values) = 0.136, 90% CI [-0.227 to 0.500], Standard Error of Mean 0.220 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 13: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M3; Test type: Superiority or Other; Mean Difference (Final Values) = 0.098, 90% CI [-0.289 to 0.485], Standard Error of Mean 0.235 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 14: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M6; Test type: Superiority or Other; Mean Difference (Final Values) = -0.202, 90% CI [-0.576 to 0.172], Standard Error of Mean 0.226 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 15: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M9; Test type: Superiority or Other; Mean Difference (Final Values) = 0.245, 90% CI [-0.180 to 0.669], Standard Error of Mean 0.257 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 16: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M12; Test type: Superiority or Other; Mean Difference (Final Values) = 0.126, 90% CI [-0.284 to 0.535], Standard Error of Mean 0.248 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 17: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M15; Test type: Superiority or Other; Mean Difference (Final Values) = 0.023, 90% CI [-0.395 to 0.441], Standard Error of Mean 0.253 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 18: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M18; Test type: Superiority or Other; Mean Difference (Final Values) = 0.146, 90% CI [-0.262 to 0.554], Standard Error of Mean 0.247 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 19: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M21; Test type: Superiority or Other; Mean Difference (Final Values) = 0.321, 90% CI [-0.138 to 0.780], Standard Error of Mean 0.278 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 20: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M24; Test type: Superiority or Other; Mean Difference (Final Values) = 0.043, 90% CI [-0.419 to 0.506], Standard Error of Mean 0.280 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 21: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M27; Test type: Superiority or Other; Mean Difference (Final Values) = 0.190, 90% CI [-0.279 to 0.659], Standard Error of Mean 0.284 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 22: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M30; Test type: Superiority or Other; Mean Difference (Final Values) = -0.117, 90% CI [-0.579 to 0.346], Standard Error of Mean 0.280 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 23: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M33; Test type: Superiority or Other; Mean Difference (Final Values) = 0.262, 90% CI [-0.189 to 0.714], Standard Error of Mean 0.273 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 24: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M36; Test type: Superiority or Other; Mean Difference (Final Values) = 0.267, 90% CI [-0.370 to 0.904], Standard Error of Mean 0.383 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height
Statistical Analysis 25: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext M36 LOCF; Test type: Superiority or Other; Mean Difference (Final Values) = 0.399, 90% CI [-0.003 to 0.802], Standard Error of Mean 0.244 — [estimate comment as in outcome 2, analysis 25]
Statistical Analysis 26: Comparison: Inhaled Insulin (Exubera®) vs Subcutaneous Insulin; Ext FU M3; Test type: Superiority or Other; Mean Difference (Final Values) = 0.619, 90% CI [0.137 to 1.102], Standard Error of Mean 0.292 — Adjusted Primary Analysis Model includes terms of treatment, baseline PFTs, center, age, sex, and height

17. Primary Outcome: Summary of ≥ 20 % Decliners in DLco
Description: Number of subjects with a post-baseline DLco decrease of ≥ 20 % [(baseline observed value - visit observed value)/(baseline observed value) * 100]; in the absence of an obvious intercurrrent illness, a repeat DLco was performed.
Time Frame: Month 3 through extension follow up Month 3
Population: FAS FEV1; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively.
Measure: Number; unit: participants
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 308 | 303
participants
  M3 (n=289, 290) | 0 | 2
  M6 (n=278, 280) | 1 | 2
  M9 (n=266, 272) | 0 | 3
  M12 (n=258, 263) | 4 | 3
  M15 (n=246, 248) | 1 | 2
  M18(n=237, 232) | 2 | 5
  M21 (n=231, 231) | 0 | 3
  M24 (n=221, 223) | 4 | 5
  FU M1 (n=247, 220) | 2 | 4
  FU M3 (n=247, 231) | 3 | 6
  FU M6 (n=241, 219) | 5 | 5
  Ext M1 (n=159, 161) | 3 | 3
  Ext M3 (n=157, 157) | 3 | 8
  Ext M6 (n=148, 157) | 4 | 6
  Ext M9 (n=143, 155) | 4 | 7
  Ext M12 (n=141, 155) | 8 | 9
  Ext M15(n=141, 142) | 4 | 6
  Ext M18 (n=132, 138) | 6 | 7
  Ext M21(n=129, 142) | 4 | 8
  Ext M24 (n=124, 130) | 5 | 7
  Ext M27(n=123, 124) | 7 | 8
  Ext M30 (n=124, 125) | 7 | 11
  Ext M33(n=98, 113) | 1 | 4
  Ext M36 (n=52, 60) | 2 | 3
  Ext FU M3 (n=118, 114) | 6 | 10

18. Secondary Outcome: Hypoglycemic Event Rates
Description: Hypoglycemic event rate; hypoglycemic event identified by characteristic symptoms of hypoglycemia with no blood glucose (BG) check with prompt resolution with food intake, SC glucagon, or intravenous (IV) glucose; characteristic symptoms with BG of 59 mg/dL (3.2 mmol/L) or less with or without symptoms. Crude event rate = total events divided by subject months (elapsed number of months a subject was in the study at each time interval).
Time Frame: Month 1 through extension Month 36
Population: as for outcome 9
Measure: Number; unit: event rate (events/subject months)
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 315 | 303
event rate (events/subject months)
  M1 (n=315, 303) | 1.63 | 1.80
  M2 (n=307, 302) | 1.40 | 1.60
  M3 (n=297, 298) | 1.22 | 1.65
  M4 (n=289, 295) | 1.10 | 1.64
  M5 (n=284, 293) | 0.95 | 1.28
  M6 (n=283, 290) | 0.98 | 1.09
  M7 (n=280, 289) | 0.80 | 1.12
  M8 (n=276, 288) | 0.82 | 0.94
  M9 (n=275, 287) | 0.71 | 0.86
  M10 (n=273, 285) | 0.72 | 0.93
  M11 (n=267, 274) | 0.68 | 0.79
  M12 (n=264, 274) | 0.72 | 0.94
  M13 (n=263, 269) | 0.71 | 0.82
  M14 (n=260, 265) | 0.62 | 0.87
  M15 (n=256, 265) | 0.64 | 0.78
  M16 (n=254, 261) | 0.68 | 0.97
  M17 (n=252, 257) | 0.53 | 0.82
  M18 (n=246, 253) | 0.61 | 0.95
  M19 (n=245, 252) | 0.59 | 0.78
  M20 (n=242, 249) | 0.62 | 0.73
  M21 (n=241, 246) | 0.57 | 0.65
  M22 (n=236, 244) | 0.44 | 0.72
  M23 (n=236, 241) | 0.41 | 0.82
  M24 (n=229, 232) | 0.45 | 0.66
  Ext M1 (n=172, 169) | 1.16 | 1.16
  Ext M2 (n=171, 169) | 1.10 | 1.33
  Ext M3 (n=169, 169) | 1.02 | 1.12
  Ext M4 (n=167, 169) | 0.87 | 1.44
  Ext M5 (n=165, 168) | 0.91 | 1.18
  Ext M6 (n=162, 167) | 0.87 | 1.20
  Ext M7 (n=161, 167) | 1.10 | 1.41
  Ext M8 (n=158, 164) | 0.82 | 1.34
  Ext M9 (n=158, 164) | 0.56 | 1.25
  Ext M10 (n=156, 164) | 0.99 | 1.11
  Ext M11 (n=153, 164) | 0.70 | 0.92
  Ext M12 (n=152, 162) | 1.26 | 1.25
  Ext M13 (n=152, 160) | 1.07 | 1.14
  Ext M14 (n=151, 159) | 0.95 | 1.01
  Ext M15 (n=149, 156) | 0.86 | 1.25
  Ext M16 (n=149, 156) | 0.99 | 1.23
  Ext M17 (n=148, 154) | 1.20 | 1.01
  Ext M18 (n=146, 154) | 1.08 | 1.05
  Ext M19 (n=143, 152) | 1.25 | 1.21
  Ext M20 (n=142, 152) | 1.20 | 1.08
  Ext M21 (n=141, 151) | 0.78 | 1.15
  Ext M22 (n=141, 149) | 0.79 | 1.08
  Ext M23 (n=139, 149) | 0.82 | 1.06
  Ext M24 (n=138, 147) | 0.88 | 1.11
  Ext M25 (n=137, 146) | 0.73 | 1.22
  Ext M26 (n=137, 145) | 0.68 | 1.25
  Ext M27 (n=137, 141) | 0.62 | 1.04
  Ext M28 (n=135, 137) | 0.68 | 0.87
  Ext M29 (n=135, 137) | 0.81 | 0.91
  Ext M30 (n=133, 137) | 0.64 | 0.87
  Ext M31 (n=124, 133) | 0.67 | 1.32
  Ext M32 (n=117, 125) | 0.82 | 0.81
  Ext M33 (n=100, 117) | 0.55 | 0.89
  Ext M34 (n=84, 90) | 0.64 | 0.57
  Ext M35 (n=66, 78) | 0.63 | 0.80
  Ext M36 (n=51, 60) | 0.72 | 0.47
  Overall comparative (n=315, 303) | 0.95 | 1.19
  Overall extension (n=172, 169) | 0.89 | 1.10

19. Secondary Outcome: Severe Hypoglycemic Event Rates
Description: Severe hypoglycemic event rate; all 3 criteria were met: subject unable to treat self, exhibited at least 1 neurological symptom (memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty awakening, suspected seizure, loss of consciousness); BG measurement ≤49 mg/dL, or not measured but clinical manifestations reversed by oral carbohydrates, SC glucagon, or IV glucose. Crude event rate: total events divided by subject months multiplied by 100 ([total events/subject months]*100). Subjects months: elapsed number of months subject was in study in each time interval.
Time Frame: Month 1 through extension Month 36
Population: as for outcome 9
Measure: Number; unit: event rate (events/subject months*100)
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 315 | 303
event rate (events/subject months*100)
  M1 (n=315, 303) | 0.98 | 0.67
  M2 (n=307, 302) | 0.34 | 0.34
  M3 (n=297, 298) | 0.69 | 0.34
  M4 (n=289, 295) | 0.35 | 1.38
  M5 (n=284, 293) | 0.36 | 1.74
  M6 (n=283, 290) | 0.72 | 2.10
  M7 (n=280, 289) | 0.00 | 0.70
  M8 (n=276, 288) | 0.37 | 0.70
  M9 (n=275, 287) | 0.74 | 0.35
  M10 (n=273, 285) | 0.00 | 0.36
  M11 (n=267, 274) | 0.38 | 0.37
  M12 (n=264, 274) | 0.76 | 0.37
  M13 (n=263, 269) | 0.77 | 0.76
  M14 (n=260, 265) | 0.78 | 0.38
  M15 (n=256, 265) | 0.79 | 0.77
  M16 (n=254, 261) | 0.00 | 0.00
  M17 (n=252, 257) | 0.00 | 0.40
  M18 (n=246, 253) | 0.00 | 0.40
  M19 (n=245, 252) | 0.41 | 0.00
  M20 (n=242, 249) | 0.42 | 0.00
  M21 (n=241, 246) | 0.00 | 0.00
  M22 (n=236, 244) | 0.00 | 0.00
  M23 (n=236, 241) | 0.00 | 0.85
  M24 (n=229, 232) | 0.00 | 0.00
  Ext M1 (n=172, 169 | 0.95 | 0.93
  Ext M2 (n=171, 169) | 0.00 | 1.87
  Ext M3 (n=169, 169) | 1.92 | 0.94
  Ext M4 (n=167, 169) | 1.92 | 0.00
  Ext M5 (n=165, 168) | 0.00 | 0.00
  Ext M6 (n=162, 167) | 0.00 | 0.94
  Ext M7 (n=161, 167) | 0.00 | 1.90
  Ext M8 (n=158, 164) | 0.00 | 0.00
  Ext M9 (n=158, 164) | 0.00 | 2.86
  Ext M10 (n=156, 164) | 0.00 | 3.81
  Ext M11 (n=153, 164) | 0.00 | 3.86
  Ext M12 (n=152, 162) | 0.98 | 3.91
  Ext M13 (n=152, 160) | 0.00 | 0.98
  Ext M14 (n=151, 159) | 0.00 | 1.96
  Ext M15 (n=149, 156) | 1.00 | 0.00
  Ext M16 (n=149, 156) | 1.00 | 1.96
  Ext M17 (n=148, 154) | 1.00 | 0.99
  Ext M18 (n=146, 154) | 1.01 | 0.00
  Ext M19 (n=143, 152) | 1.03 | 0.99
  Ext M20 (n=142, 152) | 4.16 | 0.99
  Ext M21 (n=141, 151) | 0.00 | 0.00
  Ext M22 (n=141, 149) | 0.00 | 1.00
  Ext M23 (n=139, 149) | 0.00 | 0.00
  Ext M24 (n=138, 147) | 1.06 | 2.02
  Ext M25 (n=137, 146) | 0.00 | 1.01
  Ext M26 (n=137, 145) | 0.00 | 0.00
  Ext M27 (n=137, 141) | 1.07 | 0.00
  Ext M28 (n=135, 137) | 0.00 | 0.00
  Ext M29 (n=135, 137) | 0.00 | 1.06
  Ext M30 (n=133, 137) | 0.00 | 0.00
  Ext M31 (n=124, 133) | 0.00 | 1.15
  Ext M32 (n=117, 125) | 0.00 | 3.58
  Ext M33 (n=100, 117) | 0.00 | 0.00
  Ext M34 (n=84, 90) | 0.00 | 1.89
  Ext M35 (n=66, 78) | 0.00 | 0.00
  Ext M36 (n=51, 60) | 0.00 | 0.82
  Overall comparative (n=315, 303) | 0.45 | 0.65
  Overall extension (n=172, 169) | 0.50 | 1.17

20. Secondary Outcome: Cough Questionnaire
Description: Clinician administered 6 question instrument to measure cough frequency (night, day), severity, timing in relation to short-acting insulin dosing, severity related to insulin dosing (SC or inhaled), and productivity of cough; range 0 (indicates no symptoms) to 4 (indicates severe symptoms). Questionnaire administered at Week 0 then if and only if, cough is identified as an adverse event not explained by a concomitant condition, such as an upper respiratory tract infection.
Time Frame: Week 0 and if indicated through extension follow up Month 3
Population: FAS. Due to early termination of study a limited set of analyses were undertaken and results of Cough Questionnaire were not summarized as planned.
Measure: Number; unit: scores on scale
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Baseline Dyspnea Index (BDI)
Description: Clinician administered instrument to measure the baseline severity of breathlessness (shortness of breath) in symptomatic patients with 3 domains: functional impairment, magnitude of task, and magnitude of effort. BDI score range 0 (very severe impairment) to 4 (no impairment) scaled to a BDI focal score (0-12). Lower score indicates greater impairment.
Time Frame: Week -1
Population: FAS FEV1. Due to early termination of study a limited set of analyses were undertaken and results of BDI were not summarized as planned.
Measure: Number; unit: scores on scale
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Transition Dyspnea Index (TDI)
Description: Clinician administered instrument to measure the baseline severity of breathlessness (shortness of breath) in symptomatic patients with 3 domains: functional impairment, magnitude of task, and magnitude of effort. TDI score range -3 (major deterioration) to +3 (major improvement); sum of all domains yields the TDI focal score (-9 to +9); lower score indicates greater deterioration. Compared to previous scoring to determine deterioration or improvement.
Time Frame: Week 4 through extension follow up Month 3 or end of study
Population: FAS FEV1. Due to early termination of study a limited set of analyses were undertaken and results of TDI were not summarized as planned.
Measure: Number; unit: scores on scale
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: High Resolution Computerized Tomography (HRCT) Scan: Within Normal Limits (Yes or No) at Observation When Baseline HRCT Was Within Normal Limits
Description: Number of subjects with Yes or No responses (within normal limits at specified time points = Yes or not within normal limits at specified time points = No) at observation when HRCT of thorax was within normal limits at baseline.
Time Frame: Baseline, M12, M24, Ext M6, Ext M18, Ext M36
Population: All subjects analysis substudy population: subjects from participating sites with a baseline and subsequent post-baseline HRCT measurement. Subjects were recruited prior to randomization; substudy enrollment continued until at least 50 subjects randomized to inhaled insulin were enrolled or until enrollment in the study was complete.
Measure: Number; unit: participants
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 71 | 76
participants
  M12 = Yes | 67 | 64
  M12 = No | 4 | 12
  M24 = Yes | 38 | 51
  M24 = No | 8 | 10
  Ext M6 = Yes | 32 | 37
  Ext M6 = No | 8 | 8
  Ext M18 = Yes | 28 | 33
  Ext M18 = No | 8 | 6
  Ext M36 = Yes | 22 | 27
  Ext M36 = No | 6 | 4

24. Secondary Outcome: High Resolution Computerized Tomography (HRCT) Scan: Within Normal Limits (Yes or No) at Observation When Baseline HRCT Was Not Within Normal Limits
Description: Number of subjects with Yes or No responses (within normal limits at specified time points = Yes or not within normal limits at specified time points = No) at observation when HRCT of thorax was not within normal limits at baseline. "No" response at observation further categorized as no significant change (NSC), more abnormal (> Abn), or less abnormal (< Abn).
Time Frame: Baseline, M12, M24, Ext M6, Ext M18, Ext M36
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 26 | 21
participants
  M12 = Yes | 6 | 5
  M12 = No | 20 | 16
  M12 = No (NSC) | 19 | 11
  M12 = No (> Abn) | 0 | 2
  M12 = No (< Abn) | 1 | 3
  M24 = Yes | 4 | 6
  M24 = No | 17 | 9
  M24 = No (NSC) | 17 | 8
  M24 = No (> Abn) | 0 | 1
  M24 = No (< Abn) | 0 | 0
  Ext M6 = Yes | 3 | 3
  Ext M6 = No | 16 | 9
  Ext M6 = No (NSC) | 15 | 8
  Ext M6 = No (> Abn) | 1 | 1
  Ext M6 = No (< Abn) | 0 | 0
  Ext M18 = Yes | 3 | 2
  Ext M18 = No | 14 | 7
  Ext M18 = No (NSC) | 12 | 7
  Ext M18 = No (> Abn) | 1 | 0
  Ext M18 = No (< Abn) | 1 | 0
  Ext M24 = Yes | 5 | 2
  Ext M24 = No | 9 | 8
  Ext M24 = No (NSC) | 8 | 8
  Ext M24 = No (> Abn) | 1 | 0
  Ext M24 = No (< Abn) | 0 | 0

25. Secondary Outcome: Insulin Antibodies
Description: Observed values for insulin antibodies measured as micro units per milliliter (microU/mL).
Time Frame: Baseline through extension Month 36
Population: FAS; (n)=number of subjects with analyzable data at observation: inhaled insulin/SC insulin, respectively. Insulin antibody levels increased in Exubera®-treated compared to control subjects; results are included to establish there were no safety consequences due to these elevations although this was not an originally specified protocol endpoint.
Measure: Median (Full Range); unit: microU/mL
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Number analyzed (Participants) | 312 | 300
microU/mL
  Baseline (n=312, 300) | 1.05 [1.05 to 328.00] | 1.05 [1.05 to 1077.00]
  W3 (n=270, 264) | 1.05 [1.05 to 948.00] | 1.05 [1.05 to 552.00]
  W6 (n=289, 282) | 4.40 [1.05 to 7296.00] | 1.05 [1.05 to 2123.00]
  M3 (n=293, 289) | 12.00 [1.05 to 2748.00] | 1.05 [1.05 to 4016.00]
  W18 (n=275, 280) | 18.00 [1.05 to 1051.00] | 1.05 [1.05 to 3648.00]
  M6 (n=276, 279) | 20.00 [1.05 to 1424.00] | 1.05 [1.05 to 3380.00]
  M9 (n=267, 277) | 22.00 [1.05 to 1776.00] | 1.05 [1.05 to 3412.00]
  M12 (n=263, 263) | 19.00 [1.05 to 1464.00] | 1.05 [1.05 to 1200.00]
  M15 (n=252, 253) | 20.00 [1.05 to 1760.00] | 1.05 [1.05 to 1780.00]
  M18 (n=241, 239) | 20.00 [1.05 to 1680.00] | 1.05 [1.05 to 1820.00]
  M21 (n=234, 233) | 19.00 [1.05 to 1331.00] | 1.05 [1.05 to 2230.00]
  M24 (n=226, 233) | 20.00 [1.05 to 1330.00] | 1.05 [1.05 to 1965.00]
  FU M1 (n=247, 226) | 14.00 [1.05 to 974.00] | 1.05 [1.05 to 2135.00]
  FU M3 (n=249, 229) | 8.50 [1.05 to 686.00] | 1.05 [1.05 to 1070.00]
  FU M6 (n=250, 227) | 6.55 [1.05 to 641.00] | 1.05 [1.05 to 1480.00]
  Ext M1 (n=165, 160) | 13.00 [1.05 to 894.00] | 1.05 [1.05 to 1270.00]
  Ext M3 (n=159, 158) | 15.00 [1.05 to 755.00] | 1.05 [1.05 to 765.00]
  Ext M6 (n=157, 156) | 12.00 [1.05 to 1200.00] | 1.05 [1.05 to 612.00]
  Ext M9 (n=150, 157) | 11.50 [1.05 to 1855.00] | 1.05 [1.05 to 905.00]
  Ext M12 (n=148, 154) | 13.00 [1.05 to 1535.00] | 1.05 [1.05 to 683.00]
  Ext M15 (n=144, 147) | 10.50 [1.05 to 1860.00] | 1.05 [1.05 to 770.00]
  Ext M18 (n=140, 144) | 13.00 [1.05 to 1080.00] | 1.05 [1.05 to 455.00]
  Ext M21 (n=136, 145) | 12.00 [1.05 to 801.00] | 1.05 [1.05 to 620.00]
  Ext M24 (n=130, 135) | 10.50 [1.05 to 831.00] | 1.05 [1.05 to 696.00]
  Ext M27 (n=129, 131) | 12.00 [1.05 to 885.00] | 2.50 [1.05 to 208.00]
  Ext M30 (n=125, 127) | 8.40 [1.05 to 510.00] | 1.05 [1.05 to 429.00]
  Ext M33 (n=103, 114) | 9.20 [1.05 to 700.00] | 1.05 [1.05 to 637.00]
  Ext M36 (n=56, 63) | 5.75 [1.05 to 168.00] | 1.05 [1.05 to 321.00]

ADVERSE EVENTS:
Description: Adverse events for this study are reported using MedDRA in Basic Results but are reported using COSTART in the Clinical Study Report (CSR) and PhRMA Web Synopsis (PWS) for consistency with earlier studies. Consequently, subtle differences may be observed.
Arm/Group | Inhaled Insulin (Exubera®) | Subcutaneous Insulin
Serious Adverse Events (participants affected / at risk) | 76/316 | 76/311
Other Adverse Events (participants affected / at risk) | 308/316 | 301/311
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Insulin (Exubera®) (N=316) | Subcutaneous Insulin (N=311)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarctionAcute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 1 | 3
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 5 | 3
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 4 | 5
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric volvulus (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 5
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Appendicitis (Infections and infestations) | 3 | 0
Arthritis infective (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 7 | 5
Dengue fever (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Gastritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 2
Lobar pneumonia (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 3 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3
Post procedural infection (Infections and infestations) | 1 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Device migration (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Failure of implant (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Heart rate irregular (Investigations) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cataplexy (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 0
Global amnesia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Bipolar II disorder (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Panic disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Foot amputation (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Leg amputation (Surgical and medical procedures) | 0 | 1
Shoulder operation (Surgical and medical procedures) | 0 | 1
Vascular operation (Surgical and medical procedures) | 0 | 1
Angiopathy (Vascular disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 2
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Insulin (Exubera®) (N=316) | Subcutaneous Insulin (N=311)
Abdominal pain (Gastrointestinal disorders) | 13 | 16
Diarrhoea (Gastrointestinal disorders) | 49 | 27
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19 | 15
Nausea (Gastrointestinal disorders) | 24 | 29
Vomiting (Gastrointestinal disorders) | 15 | 17
Asthenia (General disorders) | 23 | 21
Chest pain (General disorders) | 20 | 20
Fatigue (General disorders) | 19 | 30
Oedema peripheral (General disorders) | 38 | 42
Seasonal allergy (Immune system disorders) | 12 | 21
Bronchitis (Infections and infestations) | 45 | 22
Cellulitis (Infections and infestations) | 18 | 8
Gastroenteritis (Infections and infestations) | 14 | 17
Gastroenteritis viral (Infections and infestations) | 23 | 17
Influenza (Infections and infestations) | 63 | 76
Lower respiratory tract infection (Infections and infestations) | 22 | 14
Nasopharyngitis (Infections and infestations) | 83 | 94
Sinusitis (Infections and infestations) | 41 | 46
Upper respiratory tract infection (Infections and infestations) | 104 | 101
Urinary tract infection (Infections and infestations) | 29 | 30
Hyperlipidaemia (Metabolism and nutrition disorders) | 18 | 18
Hypoglycaemia (Metabolism and nutrition disorders) | 245 | 247
Arthralgia (Musculoskeletal and connective tissue disorders) | 51 | 43
Back pain (Musculoskeletal and connective tissue disorders) | 43 | 52
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 16
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 21 | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 15 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 41 | 43
Dizziness (Nervous system disorders) | 37 | 45
Headache (Nervous system disorders) | 43 | 28
Hypoaesthesia (Nervous system disorders) | 19 | 20
Tremor (Nervous system disorders) | 37 | 50
Depression (Psychiatric disorders) | 21 | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 142 | 70
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 17
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 21
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 | 29
Productive cough (Respiratory, thoracic and mediastinal disorders) | 16 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 20 | 27
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 21 | 30
Rash (Skin and subcutaneous tissue disorders) | 17 | 16
Hypertension (Vascular disorders) | 52 | 62

LIMITATIONS AND CAVEATS:
Due to early termination of study, none of the subjects completed the study as planned. Subjects active at the time of study termination completed an end-of-study assessment and a 3-month follow-up visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.